CLINICAL TRIAL: NCT02483676
Title: Adaptive Ankle Robot Control System to Reduce Foot-drop in Chronic Stroke
Brief Title: Ankle Robot to Reduce Foot Drop in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N1699-R
Record Dates: First submitted 2015-06-19; First posted 2015-06-29 (Estimated); Results first posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Stroke; Foot Drop
Keywords: Rehabilitation; Robotics; Gait
MeSH Terms: conditions — Stroke; Peroneal Neuropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treadmill+anklebot (Experimental): This group will receive gait training on a treadmill while wearing the anklebot with the adaptive control system.
  Interventions: Device: Treadmill plus anklebot
- Treadmill only (Active Comparator): This group will receive gait training on a treadmill, without use of the anklebot.
  Interventions: Behavioral: Treadmill only

INTERVENTIONS:
Device: Treadmill plus anklebot — This intervention employs the use of the adaptive anklebot control system to complement treadmill exercise training over a 6-week intervention period.
  Other Names: TMR
  Arms: Treadmill+anklebot
Behavioral: Treadmill only — This intervention employs the use of a treadmill for gait exercise training over a 6-week intervention period
  Other Names: TM
  Arms: Treadmill only

SUMMARY:
Deficits in ankle control after stroke can lead to foot drop, resulting in inefficient, aberrant gait and an elevated falls risk. Using a novel ankle robot and newly invented adaptive control system, this study tests whether robotic-assisted treadmill training will improve gait and balance functions in chronic stroke survivors with foot drop impairment. It is hypothesized that, compared to treadmill training alone, integrating adaptive ankle robotics with treadmill training will reduce drop foot during independent overground walking, resulting in greater mobility, improved postural control, and reduced fall risk.

DETAILED DESCRIPTION:
This proposal investigates a novel ankle robot (anklebot) adaptive control approach integrated with treadmill training to reduce foot drop and improve mobility function in chronic hemiparetic stroke survivors. Currently, stroke survivors with foot drop are trained to live with a cane or other assistive device, and often ankle foot orthotics (AFOs) for safety. Neither mediates task-practice or neuromotor recovery.

The investigators have developed an adaptive anklebot controller that detects gait cycle sub-events for precise timing of graded robotics assistance to enable deficit severity-adjusted ankle motor learning in the context of walking. The investigators' pilot findings show that 6 weeks treadmill training with anklebot (TMR) timed to assist swing phase dorsiflexion only is more effective than treadmill alone (TM) to improve free-walking swing dorsiflexion at foot strike, floor-walking speed, and the benefits are retained at 6 weeks post-training. Notably, swing-phase TMR training improved paretic leg push-off, and reduced center-of-pressure sway on standing balance, indicating potential benefits to other elements of gait and balance, beyond those robotically targeted toward foot drop.

This randomized study investigates the hypothesis that 6 weeks TMR is more effective to improve durably gait biomechanics, static, and dynamic balance, and mobility function in chronic stroke survivors with dorsiflexion deficits, compared to TM alone. Aims are to determine the compare effectiveness of 6 weeks TMR vs. TM alone on:

1. Independent gait function indexed by gait velocity, swing-phase DF (dorsiflexion), terminal stance push-off.
2. Balance function indexed by measures of postural sway (CoP), asymmetric loading in quiet standing, peak paretic A-P forces in non-paretic gait initiation, and standardized scales for balance and fall risk.
3. Long-term mobility outcomes, assessed by repeated measures of all key gait and balance outcomes at 6 weeks and 3 months after formal training cessation.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke > 2 months prior in men or women
* Residual hemiparesis of the lower extremity that includes symptoms of foot drop
* Capable of ambulating on a treadmill with handrail support
* Already completed all conventional physical therapy
* Adequate language and cognitive function to provide informed consent and participate in testing and training

Exclusion Criteria:

* Cardiac history of:

  * Unstable angina
  * Recent (< 3 months) myocardial infarction
  * Congestive heart failure (NYHA category II or higher)
  * Hemodynamic valvular dysfunction
  * Hypertension that is a contraindication for a bout of treadmill training (>160/100 mmHg on two assessments)
* Medical history of:

  * Recent hospitalization (< 3 months) for any serious condition leading to significant bed-rest or reduction in mobility function
  * Symptomatic peripheral arterial occlusive disease
  * Orthopedic or chronic pain conditions restricting exercise
  * Pulmonary failure requiring oxygen
  * Uncompensated renal failure
  * Active cancer
* Neurological history and exam consistent with:

  * Dementia
  * Receptive or global aphasia that confounds testing and training, operationally defined as unable to follow 2-point commands
  * Non-stroke neurological disorder restricting exercise (e.g. Parkinson's Syndrome, myopathy)
  * Untreated major depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Kittner, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treadmill+Anklebot | Treadmill Only
Started | 23 | 22
Completed | 17 | 17
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Population: 45 patients were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treadmill+Anklebot | Treadmill Only | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 15 | 12 | 27
Age, Continuous [Mean (Full Range); unit: years] | 64 [30 to 75] | 65 [30 to 75] | 65 [30 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 14 | 14 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 15 | 30
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 22 | 45
Years since stroke [Count of Participants; unit: Participants]
  <2 | 4 | 2 | 6
  2-4 | 7 | 9 | 16
  4-6 | 4 | 7 | 11
  6+ | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Gait Velocity During Self-selected Overground Walking
Description: Gait velocity during self-selected overground walking measured in cm/sec
Time Frame: Change from baseline to: Post 6-week training, 6 weeks after completion, and 3 (or 6) months after completion
Population: Only 38 of patients were included in the intention-to-treat analysis, as we excluded patients who had no baseline or follow-up data on the primary outcomes.
Measure: Mean (Standard Deviation); unit: CM/SEC
Arm/Group | Treadmill+Anklebot | Treadmill Only
Number analyzed (Participants) | 17 | 21
CM/SEC
  Baseline | 0.48 (0.21) | 0.48 (0.34)
  Post 6-week training | 0.54 (0.24) | 0.56 (0.32)
  6 weeks after completion | 0.53 (0.24) | 0.55 (0.33)
  3 (or 6) months after completion | 0.52 (0.23) | 0.55 (0.33)

2. Primary Outcome: Anterior-posterior Propulsion Forces of Paretic Side During Gait
Description: Newtons: anterior-posterior force generated during push-off phase of the gait cycle
Time Frame: Change from baseline to: Post 6-weeks training, 6 weeks after completion, and 3 (or 6) months
Population: Only 38 are included in the intention-to-treat analysis, as we excluded patients with no baseline or follow-up data on the primary outcomes.
Measure: Mean (Standard Deviation); unit: Force in Newtons
Arm/Group | Treadmill+Anklebot | Treadmill Only
Number analyzed (Participants) | 17 | 21
Force in Newtons
  Baseline | 2.22 (12.37) | 2.22 (12.37)
  Post 6-week training | 4.92 (10.99) | 3.03 (10.99)
  6 weeks after completion | 6.06 (8.92) | 4.14 (8.92)
  3 (or 6) months after completion | 4.88 (10.74) | 3.98 (10.74)

3. Primary Outcome: Peak Dorsiflexion Angle During Swing Phase of Gait
Description: Degrees; extent of ankle dorsiflexion to enable foot clearance
Time Frame: Change from baseline to: Post 6-week training, 6 weeks after completion, and 3 (or 6) months after completion
Population: Only 38 are included in the intention-to-treat analysis, as we excluded patients who had no baseline or follow-up data on the primary outcomes.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Treadmill+Anklebot | Treadmill Only
Number analyzed (Participants) | 17 | 21
Degrees
  Baseline | 3.95 (6.83) | 3.95 (6.83)
  Post 6-week training | 4.84 (6.83) | 4.24 (6.83)
  6 weeks after completion | 4.34 (6.26) | 3.27 (6.26)
  3 (or 6) months after completion | 3.33 (6.72) | 3.43 (6.72)

4. Primary Outcome: Postural Sway Areas During Quiet Standing
Description: cm^2; extent of postural deviations to assess static postural control
Time Frame: Change from baseline to: Post 6-week training, 6 weeks after completion, and 3 (or 6) months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: CM^2
Arm/Group | Treadmill+Anklebot | Treadmill Only
Number analyzed (Participants) | 17 | 21
CM^2
  Baseline | 1.16 (0.64) | 1.16 (0.64)
  Post 6-week training | 1.51 (0.82) | 1.33 (0.82)
  6 weeks after completion | 1.44 (0.57) | 1.13 (0.52)
  3 (or 6) months after completion | 1.59 (0.52) | 1.14 (0.52)

5. Primary Outcome: Ratio of Asymmetric Loading in Quiet Standing
Description: Ratio of Newtons of force per each leg (paretic/nonparetic) while standing quietly
Time Frame: Change from baseline to: Post 6-week training, 6 weeks after completion, and 3 (or 6) months
Population: This data was not recorded during the study nor calculated as part of the analysis.
Arm/Group | Treadmill+Anklebot | Treadmill Only
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Peak Paretic Push Off Forces During Gait Initiation
Description: Newtons; magnitude of forward ground reaction forces
Time Frame: Change from baseline to: Post 6-week training, 6 weeks after completion, and 3 (or 6) months
Population: Only 38 are included in the intention-to-treat analysis, as we excluded patients who had no baseline or follow-up data on the primary outcomes.
  The results should be interpreted with extreme caution as there was inconsistent use of AFO's (ankle-foot orthosis) during evaluations and/or the training focus was on dorsiflexion assistance.
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | Treadmill+Anklebot | Treadmill Only
Number analyzed (Participants) | 17 | 21
Newtons
  Baseline | 64.7 (28.5) | 64.7 (28.5)
  Post 6-week training | 63.5 (27) | 62.8 (27)
  6 weeks after completion | 65.4 (30.6) | 69.8 (30.6)
  3 (or 6) months after completion | 66.1 (29.9) | 70.9 (29.9)

7. Post Hoc Outcome: Dorsiflexion Angle at Foot Strike
Description: Degrees, extent of ankle dorsiflexion at initial foot contact with the floor
Time Frame: Change from baseline to: Post 6-week training, 6 weeks after completion, and 3 (or 6) months after completion
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Treadmill+Anklebot | Treadmill Only
Number analyzed (Participants) | 17 | 21
Degrees
  Baseline | -1.83 (5.03) | -1.83 (7.31)
  Post 6-week training | -0.70 (6.55) | -0.46 (5.7)
  6 weeks after completion | -2.18 (6.27) | -2.15 (6.16)
  3 (or 6) months after completion | -2.99 (5.96) | -1.58 (6.71)

ADVERSE EVENTS:
Time Frame: 24 to 36 weeks for each subject; 6 week training + 6 weeks post training + 12 or 24 weeks follow up
Arm/Group | Treadmill+Anklebot | Treadmill Only
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 4/23 | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treadmill+Anklebot (N=23) | Treadmill Only (N=22)
Pre-existing Medical Condition (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Knee pain
Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Leg soreness, foot swelling
Weakness (Cardiac disorders) | 0 (0) | 2 (2) — Dizziness, weakness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT02483676/SAP_001.pdf
  • Informed Consent Form (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT02483676/ICF_002.pdf
  • Study Protocol (2015-05-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT02483676/Prot_003.pdf